CLINICAL TRIAL: NCT02723812
Title: A Bridging Study to Evaluate Safety of GCFLU® One Dose (0.5ml) (Seasonal Influenza Vaccine) Administered Intramuscularly in Healthy Vietnamese Volunteer Aged From 3 Years Old
Brief Title: Evaluate Safety of GCFLU® Administered Intramuscularly in Healthy Vietnamese Volunteer Aged From 3 Years Old
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Clinical Research and Clinical Trial Support for Vaccine and Biological Products (Other)
Collaborators: Green Cross Corporation (Industry)
Responsible Party: Principal Investigator, Nguyen Vu Thuong, Vice Director, Pasteur Institute, Ho Chi Minh City
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VX-2015.02
Record Dates: First submitted 2016-02-22; First posted 2016-03-30 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Influenza, Human
Keywords: Influenza; GCFLU; vaccine; Vietnam
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GCFLU® Influenza vaccine (Split virion, Inactivated) (Experimental): One dose 0.5 mL vaccine GCFLU® administered intramuscularly.
  Interventions: Biological: GCFLU® Influenza vaccine (Split virion, Inactivated)

INTERVENTIONS:
Biological: GCFLU® Influenza vaccine (Split virion, Inactivated)
  Other Names: GCFLU® pre-filled syringe inj.

SUMMARY:
An open label, non-comparative bridging study to evaluate the safety of GCFLU® (seasonal influenza vaccine) administered intramuscularly in healthy Vietnamese volunteer aged from 3 years old

DETAILED DESCRIPTION:
A bridging study to evaluate safety of seasonal influenza vaccine GCFLU® pre-filled syringe inj. One dose (0.5 ml) after exposure administered intramuscularly. The study conducted in Ben Luc District of Long An province, in which 120 healthy Vietnamese volunteer aged from 5 year old will be enroll to the study. All subject will receive only one dose (0.5 ml) vaccine in Day 0.

Study variables will be collected to determine and provide the evidence for the safety of GCFLU®, include:

* Local and systemic adverse event (AE) in 30 minutes after vaccination.
* Local and systemic AE in 7 days after vaccination
* Unsolicited AE over 21 days after vaccination.
* Serious adverse event (SAE) after vaccination and in 21 days of observation periods Study protocol has been reviewed and approved by Pasteur Institute in Ho Chi Minh City (HCMC) Institutional Review Board (IRB), Vietnam Ministry of Health - Independent Ethics Committee (IEC) and Vietnam Minister of Health.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all criteria below to participate in study

1. A person who is a 3-year-old or older, healthy and can be followed up for 21 days
2. Subject who gave voluntary written consent to participate in the study, and able to comply with the study requirements. With subjects aged from 3 years to below 18 years, parents/legal representative will give voluntary consent to participate in this study, and subjects from 12 to under 18 years old will give voluntary written consent for children.

Exclusion Criteria:

Subject have one of criteria below must not participate in study

1. Subject with a known hypersensitivity or allergic reaction to eggs or eggs products, to chicken or chicken products, to any component of the study vaccine, neomycin or gentamicin.
2. Subjects with immune system disorder including immune deficiency disease.
3. Subjects with a history of Guillain-Barre syndrome.
4. Subjects with severe chronic disease (e.g.; cardiovascular disease except for controlled hypertension, respiratory disease, metabolic disease, renal/kidney dysfunction or hemoglobinopathy etc.) who in the investigator's opinion may have a difficulty in participating in the study.
5. Subjects with hemophilia or receiving a treatment with an anticoagulant, who are at increased risk of serious bleeding during intramuscular injection.
6. Subject who had acute fever with body temperature exceeding 37.50 Celsius (armpit calculated) before vaccination with the study drug.
7. Subjects who had received other vaccination within 14 days before vaccination with the study drug, or those who had another vaccination scheduled during the study.
8. Pregnant women, breast-feeding women or women of childbearing potential who do not use an appropriate method of contraception (use of condom, intrauterine contraceptive device, or hormone contraceptives, or of a male partner had vasectomy).
9. Subjects who had participated in other clinical study within 28 days priors to vaccination with the study drug, or those who had another clinical trial scheduled during the study.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Safety of GCFLU® by assessing the frequency, rate and severity of adverse events (local and general). | 30 minutes after vaccination.
Safety of GCFLU® by assessing the frequency, rate and severity of solicited adverse events (local and general) | For 7 days after vaccination.
Safety of GCFLU® by assessing the frequency, rate and severity of unsolicited adverse events. | During 21 days after vaccination.
Safety of GCFLU® by assessing the frequency, rate and severity of serious adverse events. | During 21 days after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Thuong Nguyen Vu, PhD., Principal Investigator — Pasteur Institute, Ho Chi Minh City
Locations (1):
- Ben Luc Health centre, Bến Lức, Long An, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided